CLINICAL TRIAL: NCT05449886
Title: Study on the Prediction of Fluid Responsiveness in Pediatric Patients Undergoing General Anesthesia With Prone Position
Brief Title: Prone Fluid Responsiveness in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2204-171-1321
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tidal volume challenge (Experimental)
  Interventions: Procedure: TVC

INTERVENTIONS:
Procedure: TVC — Tidal volume challenge from 6ml/kg to 10ml/kg for 1 min.

SUMMARY:
In pediatric patients in the prone position, the reliability of pulse pressure variation and stroke volume variation, and pleth variability index to predict fluid responsiveness have not previously been established. Perioperatively, in this setting, optimizing fluid management can be challenging, and fluid overload is associated with both intraoperative and postoperative complications. The investigator designed this study to assess the sensitivity and specificity of baseline PPV, SVV, and PVI the tidal volume (VT) challenge (VTC) and in predicting fluid responsiveness during elective neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* elective neurosurgery and requiring prone positioning

Exclusion Criteria:

* (1) chronic cardiac arrhythmia; (2) depressed left (<30% of ejection fraction) (3) patients with pulmonary disease

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-12 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
fluid responsiveness prediction using AUC of ROC curve analysis | from induction of anesthesia to end of operation, about 5 hours
  stroke volume index increase more than 10% from baseline after volume administration (10ml/kg) Fluid responsiveness parameters; PPV, SVV, PVI, rPVI before and after tidal volume challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, South Korea